CLINICAL TRIAL: NCT06715384
Title: Performance Evaluation of a Computer-aided Measuring System for Colorectal Polyp Size Measurement: a Prospective Study
Brief Title: Evaluation of a CAM System for Colorectal Polyp Size Measurement
Acronym: CAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology Dept and Digestive Endoscopy Center, Changhai Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: CHEC2024-389
Record Dates: First submitted 2024-11-26; First posted 2024-12-04 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Polyp; Colorectal Adenoma
Keywords: Artificial Intelligence; Polyp Size; Deep Learning; Colonoscopy; Depth Map

STUDY DESIGN:
Intervention Model Description: prospective, multi-endoscopist, single-center or multi- centers
Who Masked: Participant
Masking Description: Randomization will be concealed. The patient will be blind to the assigned groups. The endoscopist will be blind to the allocated groups until the polyp is identified.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Polyp size measurement with Artificial intelligence (AI) (Experimental): Colonoscopies will be performed according to the standard of care. Patients will have colonoscopies performed using the computer-aided measuring (CAM) system. All measured fresh polyp specimens will be immediately sized in vitro as the ground truth.
  Interventions: Diagnostic Test: Polyp size measurement using autonomous AI measurement or AI-assisted human measurement with the CAM system
- Polyp size measurement without AI (No Intervention): Colonoscopies will be performed according to the standard of care without the CAM system. Patients will undergo a standard colonoscopy. Polyp size measurement will be assessed visually and non-scaled device (open biopsy forceps or snare). All measured fresh polyp specimens will be immediately sized in vitro as the ground truth.

INTERVENTIONS:
Diagnostic Test: Polyp size measurement using autonomous AI measurement or AI-assisted human measurement with the CAM system — The study of real-time polyp size measurement using the CAM system will be conducted in two phases. Phase I (pilot phase, n=24 polyps, about 27 patients) will be used to assess the feasibility of applying the CAM system in real-time in a clinical video in order to obtain pilot data on the relative accuracy of assessing polyp sizes using autonomous AI measurement and AI-assisted human measurement and to determine the relative accuracy of assessing polyp size in Phase II of the study ( Randomized Controlled Trial) to assess the sample size and reference standards for the CAM system. The sample size for the second phase of the randomized controlled trial (comparing AI-assisted human measurement to non-scaled device) will be based on pilot data in order to compare the relative accuracy of polyp size measurement with AI-assisted human measurement versus non-scaled device in clinical practice.
  Other Names: Polyp size measurement with the CAM system
  Arms: Polyp size measurement with Artificial intelligence (AI)

SUMMARY:
Accurate polyp size measurements are essential for risk stratification, selection of polypectomy techniques, and surveillance interval assignments. Evidence indicated that the clinical implementation of artificial intelligence is an optimal tool to improve the measurement of polyps during colonoscopy. This study aimed to evaluate the performance of a computer-aided measuring (CAM) system (EndoDASS) and compare its accuracy with routine sizing methods during real-time colonoscopy.

DETAILED DESCRIPTION:
This study will be conducted in 2 phases: the first phase will evaluate the value of the application of the computer-aided measuring (CAM) system for polyp size measurement accuracy in a small sample of clinical videos, recording the corresponding clinical videos for CAM measurements after measuring polyp size using real-time visual assessment and non-scaled device (open biopsy forceps or snare) assessment, and comparing the different methods of polyp size measurement through a video-based analysis [Autonomous artificial intelligence (AI) measurement, AI-assisted human measurement, non-scaled device assessment, and visual assessment] with different groups of endoscopists ( experts, gastroenterologists, surgeons, fellows) evaluating the corresponding clinical videos during real-time measurements, to obtain pilot data on the relative accuracy of polyp size measurement when using the CAM system, to test the feasibility of size measurement of freshly resected polyp specimens and to determine the sample size and reference for evaluating the CAM system in the subsequent phases of a randomized controlled trial of the study. The second phase will assess the value of using the AI-assisted human measurement versus the non-scaled device assessment for polyp size measurement accuracy in a clinical randomized controlled trial using a prospective, multicenter, patient-single-blind, randomized controlled trial design in which subjects are randomly assigned to the CAM group and the non-scaled device measurement group in a 1:1 ratio. Each patient will have a maximum of 3 polyps included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-75, any gender; 76-85 years eligible case-by-case based on health status.
2. Colonoscopy screening, surveillance, or diagnostic participants.
3. Informed consent obtained.

Exclusion Criteria:

1. Anticoagulant use (e.g., aspirin, warfarin) within 7 days prior to colonoscopy or coagulopathy.
2. Inflammatory bowel disease.
3. Aronchick score >3 at entry.
4. Incomplete Case Report Form (CRF) data.
5. Emergency colonoscopy.
6. Pregnancy or lactation.
7. Gastrointestinal obstruction.
8. Refusal to participate.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the computer-aided measuring (CAM) system | 7 days
  To evaluate the relative accuracies of the computer-aided measuring (CAM) system measurement (Autonomous AI measurement and AI-assisted human measurement), non-scaled device (open biopsy forceps or snare) assessment or visual assessment for measuring polyp size compared to with measurement of freshly resected polyp specimens by a digital vernier caliper as reference standard. Relative accuracy is defined as "[1-(CAM system measurement - ground truth measurement)/ground truth measurement] x100%". Scale: 0-100. Higher score is a better outcome.

SECONDARY OUTCOMES:
video-based analysis | 7 days
  Compare in video-based analysis with different endoscopists (experts, gastroenterologists, surgeons, fellows) the relative size measurements accuracy of CAM system measurement with visual and non-scaled device assessment. Relative accuracy is deﬁned as "[1-(CAM system measurement ground truth measurement)/ground truth measurement] x100%". Scale: 0-100. Higher score is a better outcome.
Reliability between CAM system measurement and ground truth measurement | 7 days
  Reliability between CAM system measurement, non-scaled device assessment, visual assessment and ground truth measurement is evaluate by concordance correlation coefficient (CCC). CCC is a statistical measure used to evaluate the agreement between two continuous variables.The CCC considers both the correlation and the bias between the two variables. It ranges from -1 to 1；1: Perfect agreement. 0: No agreement. Negative values: Indicate that the variables diverge.
Time taken for polyp size measurement | 7 days
  Measurement time of the AI-assisted human measurement, non-scaled device assessment, and visual estimation refers to the time taken by endoscopists using various measurement methods, starting from when a polyp appears in the field of view for measurement until the report of the polyp size is completed.
Percentage differences between the AI-assisted human measurement and non-scaled device assessment | 7 days
  Calculate percentage differences between the AI-assisted human measurement and non-scaled device assessment.
Instances of overestimation or underestimation by the AI-assisted human measurement and non-scaled device assessment | 7 days
  Evaluate the instances of overestimation or underestimation by the AI-assisted human measurement and non-scaled device assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Bing Zhao, MD, Principal Investigator — Department of Gastroenterology, National Clinical Research Center for Digestive Diseases, Changhai Hospital, Naval Medical University, Shanghai 200433, China.; Yu Bai, MD, Study Director — Department of Gastroenterology, National Clinical Research Center for Digestive Diseases, Changhai Hospital, Naval Medical University, Shanghai 200433, China.; En-Da Yu, MBBS, Study Director — Department of Colorectal Surgery and Gastrointestinal Endoscopy Center, Changhai hospital, Naval Medical University, Shanghai 200433, China.; Zhao-Shen Li, MD, PhD, Study Chair — Department of Gastroenterology, National Clinical Research Center for Digestive Diseases, Changhai Hospital, Naval Medical University, Shanghai 200433, China.
Locations (1):
- Changhai Hospital, Naval Medical University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
IPD data can be shared with investigators who propose to use the data under the approval of an independent review committee. Data can only be used for the goals specified in the proposal. Data sharing will be implemented between 6-18 months after article publication with a data-sharing agreement signed. Yu Bai can be contacted at the corresponding email.

REFERENCES:
- [Background] Siegel RL, Giaquinto AN, Jemal A. Cancer statistics, 2024. CA Cancer J Clin. 2024 Jan-Feb;74(1):12-49. doi: 10.3322/caac.21820. Epub 2024 Jan 17. PMID 38230766
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Wang J, Chen X, Wu L, et al. An artificial intelligence-based system for measuring the size of gastrointestinal lesions under endoscopy (with video). Chinese Journal of Digestive Endoscopy. 2022;39(12):965-971.
- [Background] Wu Y, Shih FY, Wang C, et al. The Deep Hybrid Neural Network and an Application on Polyp Detection. Intern J Pattern Recognit Artif Intell. 2024;38(04).
- [Background] Wang J, Li Y, Chen B, Cheng D, Liao F, Tan T, Xu Q, Liu Z, Huang Y, Zhu C, Cao W, Yao L, Wu Z, Wu L, Zhang C, Xiao B, Xu M, Liu J, Li S, Yu H. A real-time deep learning-based system for colorectal polyp size estimation by white-light endoscopy: development and multicenter prospective validation. Endoscopy. 2024 Apr;56(4):260-270. doi: 10.1055/a-2189-7036. Epub 2023 Oct 12. PMID 37827513
- [Background] Abdelrahim M, Saiga H, Maeda N, Hossain E, Ikeda H, Bhandari P. Automated sizing of colorectal polyps using computer vision. Gut. 2022 Jan;71(1):7-9. doi: 10.1136/gutjnl-2021-324510. Epub 2021 Jul 15. No abstract available. PMID 34266967
- [Background] Djinbachian R, Haumesser C, Taghiakbari M, Pohl H, Barkun A, Sidani S, Liu Chen Kiow J, Panzini B, Bouchard S, Deslandres E, Alj A, von Renteln D. Autonomous Artificial Intelligence vs Artificial Intelligence-Assisted Human Optical Diagnosis of Colorectal Polyps: A Randomized Controlled Trial. Gastroenterology. 2024 Jul;167(2):392-399.e2. doi: 10.1053/j.gastro.2024.01.044. Epub 2024 Feb 7. PMID 38331204
- [Background] Liu Y, Zuo S. Self-supervised monocular depth estimation for gastrointestinal endoscopy. Comput Methods Programs Biomed. 2023 Aug;238:107619. doi: 10.1016/j.cmpb.2023.107619. Epub 2023 May 19. PMID 37235969
- [Background] Su R, Liu J, Wu B, Xie Y, Zhang Y, Zhang W, Zhang Y, Wan M, Tian Z, Hu Y. Accurate measurement of colorectal polyps using computer-aided analysis. Eur J Gastroenterol Hepatol. 2021 May 1;33(5):701-708. doi: 10.1097/MEG.0000000000002162. PMID 33787542
- [Background] Zuo W, Dai Y, Huang X, Peng RQ, Li X, Liu H. Evaluation of the competence of an artificial intelligence-assisted colonoscopy system in clinical practice: A post hoc analysis. Front Med (Lausanne). 2023 Apr 6;10:1158574. doi: 10.3389/fmed.2023.1158574. eCollection 2023. PMID 37089592
- [Background] Sudarevic B, Sodmann P, Kafetzis I, Troya J, Lux TJ, Sassmannshausen Z, Herlod K, Schmidt SA, Brand M, Schottker K, Zoller WG, Meining A, Hann A. Artificial intelligence-based polyp size measurement in gastrointestinal endoscopy using the auxiliary waterjet as a reference. Endoscopy. 2023 Sep;55(9):871-876. doi: 10.1055/a-2077-7398. Epub 2023 Apr 20. PMID 37080235
- [Background] Kwak MS, Cha JM, Jeon JW, Yoon JY, Park JW. Artificial intelligence-based measurement outperforms current methods for colorectal polyp size measurement. Dig Endosc. 2022 Sep;34(6):1188-1195. doi: 10.1111/den.14318. Epub 2022 May 19. PMID 35385184
- [Background] Plumb AA, Nickerson C, Wooldrage K, Bassett P, Taylor SA, Altman D, Atkin W, Halligan S. Terminal digit preference biases polyp size measurements at endoscopy, computed tomographic colonography, and histopathology. Endoscopy. 2016 Oct;48(10):899-908. doi: 10.1055/s-0042-108727. Epub 2016 Jul 21. PMID 27441685
- [Background] Ahmad I, Levine JB, Anderson JC. Endoscopic Measurement of Colorectal Polyps: How Do We Measure Up? Gastroenterology. 2016 Mar;150(3):769-71. doi: 10.1053/j.gastro.2016.01.020. Epub 2016 Jan 25. No abstract available. PMID 26820916
- [Background] Eichenseer PJ, Dhanekula R, Jakate S, Mobarhan S, Melson JE. Endoscopic mis-sizing of polyps changes colorectal cancer surveillance recommendations. Dis Colon Rectum. 2013 Mar;56(3):315-21. doi: 10.1097/DCR.0b013e31826dd138. PMID 23392145
- [Background] Taylor JL, Coleman HG, Gray RT, Kelly PJ, Cameron RI, O'Neill CJ, Shah RM, Owen TA, Dickey W, Loughrey MB. A comparison of endoscopy versus pathology sizing of colorectal adenomas and potential implications for surveillance colonoscopy. Gastrointest Endosc. 2016 Aug;84(2):341-51. doi: 10.1016/j.gie.2016.04.009. Epub 2016 Apr 19. PMID 27102832
- [Background] Anderson BW, Smyrk TC, Anderson KS, Mahoney DW, Devens ME, Sweetser SR, Kisiel JB, Ahlquist DA. Endoscopic overestimation of colorectal polyp size. Gastrointest Endosc. 2016 Jan;83(1):201-8. doi: 10.1016/j.gie.2015.06.058. Epub 2015 Aug 28. PMID 26318830
- [Background] Taghiakbari M, Djinbachian R, Haumesser C, Sidani S, Chen Kiow JL, Panzini B, von Renteln D. Measuring Size of Colorectal Polyps Using a Virtual Scale Endoscope or Visual Assessment: A Randomized Controlled Trial. Am J Gastroenterol. 2024 Jul 1;119(7):1309-1317. doi: 10.14309/ajg.0000000000002623. Epub 2023 Dec 12. PMID 38084850
- [Background] Djinbachian R, Taghiakbari M, Haumesser C, Zarandi-Nowroozi M, Khalil MA, Sidani S, Liu J, Panzini B, von Renteln D. Comparing size measurement of colorectal polyps using a novel virtual scale endoscope, endoscopic ruler or forceps: A preclinical randomized trial. Endosc Int Open. 2023 Jan 30;11(1):E128-E135. doi: 10.1055/a-2005-7548. eCollection 2023 Jan. PMID 36726860
- [Background] von Renteln D, Djinbachian R, Zarandi-Nowroozi M, Taghiakbari M. Measuring size of smaller colorectal polyps using a virtual scale function during endoscopies. Gut. 2023 Mar;72(3):417-420. doi: 10.1136/gutjnl-2022-328654. Epub 2022 Nov 21. No abstract available. PMID 36411028
- [Background] Visentini-Scarzanella M, Kawasaki H, Furukawa R, Bonino MA, Arolfo S, Lo Secco G, Arezzo A, Menciassi A, Dario P, Ciuti G. A structured light laser probe for gastrointestinal polyp size measurement: a preliminary comparative study. Endosc Int Open. 2018 May;6(5):E602-E609. doi: 10.1055/a-0577-2798. Epub 2018 May 8. PMID 29756018
- [Background] Kaz AM, Anwar A, O'Neill DR, Dominitz JA. Use of a novel polyp "ruler snare" improves estimation of colon polyp size. Gastrointest Endosc. 2016 Apr;83(4):812-6. doi: 10.1016/j.gie.2015.08.082. Epub 2015 Sep 14. PMID 26382052
- [Background] Hyun YS, Han DS, Bae JH, Park HS, Eun CS. Graduated injection needles and snares for polypectomy are useful for measuring colorectal polyp size. Dig Liver Dis. 2011 May;43(5):391-4. doi: 10.1016/j.dld.2010.12.015. Epub 2011 Feb 21. PMID 21334993
- [Background] Kume K, Watanabe T, Yoshikawa I, Harada M. Endoscopic measurement of polyp size using a novel calibrated hood. Gastroenterol Res Pract. 2014;2014:714294. doi: 10.1155/2014/714294. Epub 2014 Jun 30. PMID 25093021
- [Background] Mir FA, Boumitri C, Ashraf I, Matteson-Kome ML, Nguyen DL, Puli SR, Bechtold ML. Cap-assisted colonoscopy versus standard colonoscopy: is the cap beneficial? A meta-analysis of randomized controlled trials. Ann Gastroenterol. 2017;30(6):640-648. doi: 10.20524/aog.2017.0180. Epub 2017 Jul 24. PMID 29118558
- [Background] Leng Q, Jin HY. Measurement system that improves the accuracy of polyp size determined at colonoscopy. World J Gastroenterol. 2015 Feb 21;21(7):2178-82. doi: 10.3748/wjg.v21.i7.2178. PMID 25717254
- [Background] Jin HY, Leng Q. Use of disposable graduated biopsy forceps improves accuracy of polyp size measurements during endoscopy. World J Gastroenterol. 2015 Jan 14;21(2):623-8. doi: 10.3748/wjg.v21.i2.623. PMID 25605986
- [Background] Rex DK, Rabinovitz R. Variable interpretation of polyp size by using open forceps by experienced colonoscopists. Gastrointest Endosc. 2014 Mar;79(3):402-7. doi: 10.1016/j.gie.2013.08.030. Epub 2013 Oct 8. PMID 24119506
- [Background] Hassan C, Antonelli G, Dumonceau JM, Regula J, Bretthauer M, Chaussade S, Dekker E, Ferlitsch M, Gimeno-Garcia A, Jover R, Kalager M, Pellise M, Pox C, Ricciardiello L, Rutter M, Helsingen LM, Bleijenberg A, Senore C, van Hooft JE, Dinis-Ribeiro M, Quintero E. Post-polypectomy colonoscopy surveillance: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2020. Endoscopy. 2020 Aug;52(8):687-700. doi: 10.1055/a-1185-3109. Epub 2020 Jun 22. PMID 32572858
- [Background] Zessner-Spitzenberg J, Waldmann E, Rockenbauer LM, Demschik A, Penz D, Trauner M, Ferlitsch M. Polyp size is associated with colorectal cancer death across histologic polyp subtypes: a retrospective study of a screening colonoscopy registry. Endoscopy. 2024 Nov;56(11):820-827. doi: 10.1055/a-2339-0146. Epub 2024 Jun 27. PMID 38936414
- [Background] Wang Y, Huang Y, Chase RC, Li T, Ramai D, Li S, Huang X, Antwi SO, Keaveny AP, Pang M. Global Burden of Digestive Diseases: A Systematic Analysis of the Global Burden of Diseases Study, 1990 to 2019. Gastroenterology. 2023 Sep;165(3):773-783.e15. doi: 10.1053/j.gastro.2023.05.050. Epub 2023 Jun 9. PMID 37302558
- [Background] Mori Y. New horizons in polyp size estimation. Endoscopy. 2024 Apr;56(4):271-272. doi: 10.1055/a-2224-0756. Epub 2024 Jan 12. No abstract available. PMID 38216131